CLINICAL TRIAL: NCT06220188
Title: [177Lu]Lu-PSMAI&T Radioligand Therapy (PSMA-RLT) for Patients With Prostate Cancer and Biochemical But Not Radio-morphological Local Recurrence After Primary Therapy With Curative Intent: A Prospective Phase II Pilot Study
Brief Title: PSMA-RLT in Biochemically Recurrent PCa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sazan Rasul, MD, PhD, Physician and post-doctoral researcher, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1938/2022; 2022-003713-11 (EudraCT Number)
Record Dates: First submitted 2023-12-25; First posted 2024-01-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer Recurrent
Keywords: [177Lu]Lu-PSMA I&T; PSMA-radioligand therapy; Biochemical recurrence; Prostate cancer; PSA value
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective single-center one-arm phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biochemical recurrent prostate cancer but not radio-morphological local recurrence (Experimental): Patients with prostate cancer and confirmed biochemical recurrence with PSA of ≥ 0.2 ng/ml after radical prostatectomy or PSA > nadir + 2ng/ml after radiotherapy but not radio-morphological local recurrence after primary therapy with curative intent will receive systemic therapy with [177Lu]Lu-PSMAI&T radioligand therapy
  Interventions: Drug: [177Lu]Lu-PSMA I&T

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA I&T — 2 cycles (3 GBq in first cycle and 6 GBq in the second cycle) of [177Lu]Lu-PSMAI&T radioligand therapy at 6-week intervals
  Other Names: PSMA-RLT

SUMMARY:
Prospective single-center one-arm phase II study in patients with prostate cancer and confirmed biochemical recurrence (BCR) with PSA of ≥ 0.2 ng/ml after radical prostatectomy (RP) or PSA > nadir + 2ng/ml after radiotherapy (RT) but not radio-morphological local recurrence after primary therapy with curative intent receive systemic therapy with only 2 cycles of highly standardized (3 GBq in first cycle and 6 GBq in the second cycle) PSMA-RLT at 6-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biochemical recurrence after radical prostatectomy and radiotherapy with a PSA doubling-time (DT) of ≤ 12 months.
* No hormonal therapy within the last 12 months or recovered testosterone levels.
* PSMA PET negative result for local recurrence; presence of distant metastases is allowed: (cN0, cM0/cM1).
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* Patients must have adequate bone marrow reserve: WBC ≥1.5 x 109 /L, Platelets ≥100 x 109 /L and Haemoglobin ≥9 g/dL.
* Patients must have adequate renal function with eGFR ≥ 50mL/min/1.73m2 using the Modification of Diet Renal Disease (MDRD) equation and an Albumin level of ≥2.5 g/dL.
* Patients must be able to sign Informed Consent Form.

Exclusion Criteria:

* Concomitant participation in any other interventional trial.
* Concurrent severe oncological and medical conditions that result in patients not having a life expectancy of longer than one year.
* Presence of clinically relevant somatic or psychiatric diseases that might interfere with the objectives and assessments of the study.
* Complete urinary out-flow obstruction or severe unmanageable urinary incontinence.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
PSA response | 12 months
  in term of PSA decline of ≥ 50% from baseline value
Emergence of therapy toxicity | 12 months
  in terms of pathological (Grade 3) reduction of values of blood count (hemoglobin decreased <8.0 g/dL; <4.9 mmol/L; <80 g/L; platelet count decreased <50,000 - 25,000/mm3; <50.0 - 25.0 x 10e9 /L and white blood cell decreased <2000 - 1000/mm3; <2.0 - 1.0 x 10e9 /L. ), kidney (creatinine increased > 3.0 x baseline or >3.0 - 6.0 x upper limit of normal (UNL)) and liver functions (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and GGT increased >5.0 - 20.0 x ULN if baseline was normal or >5.0 - 20.0 x baseline if baseline was abnormal; albumin <2 g/dL or <20 g/L; bilirubin increased >3.0 - 10.0 x ULN if baseline was normal or >3.0 - 10.0 x baseline if baseline was abnormal and lactate dehydrogenase increased > ULN.), assessed by Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Time to PSA value progression | 18 months
  to evaluate progression free survival
androgen deprivation therapy- and other treatment-free survival | 18 months
  analyze the time until the start of androgen deprivation therapy
Evaluation of life quality of the treated patients | 18 months
  Using the questionnaires: FACT-P, EORTC QLQ
Assess time to imaging progression | 18 months
  In terms of appearance of new PSMA-avid lesions and/or size progression of the metastatic lymph nodes evaluated based on response evaluation criteria of solid tumor (RECIST) version 1.1.
Quantification of circulating free tumor DNA | 18 months
  Quantification of circulating free tumor DNA (ctDNA), enumeration of circulating tumor cells (CTCs) before and following [177Lu]Lu-PSMAI&T-RLT and analyse molecular changes in liquid biopsy markers following [177Lu]Lu-PSMAI&T-RLT.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided